CLINICAL TRIAL: NCT04025073
Title: The Impact of Dietary Habits and Nutrition Intervention on Metabolic Syndrome Parameters in Hospitalized Individuals With the Diagnosis of Schizophrenia
Brief Title: The Impact of Dietary Habits and Nutrition Intervention on Metabolic Syndrome in Individuals With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tamara Sorić (Individual)
Collaborators: University of Zagreb (Other)
Responsible Party: Sponsor-Investigator, Tamara Sorić, Head of Nutrition Department, Psychiatric Hospital Ugljan
Organization: Psychiatric Hospital Ugljan (Individual)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TS_01/17
Record Dates: First submitted 2019-07-14; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Schizophrenia; Nutrition Therapy
MeSH Terms: conditions — Metabolic Syndrome; Schizophrenia | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will be assigned to the DASH diet with moderately reduced caloric intake and will participate in a nutrition education program.
  Interventions: Other: Dietary Approaches to Stop Hypertension; Other: Nutrition education program
- Control Group (Experimental): The control group will continue to follow the standard hospital diet and will participate in the same nutrition education program as the intervention group.
  Interventions: Other: Nutrition education program

INTERVENTIONS:
Other: Dietary Approaches to Stop Hypertension — The DASH diet will have a reduced caloric intake by 400 kcal/day, when compared to the standard hospital diet. The DASH diet will be planned according to the following: total daily energy intake 1,900 kcal; total daily fat intake 27%; daily intake of saturated fatty acids 6%; total daily protein intake 18%; total daily carbohydrates intake 55%; cholesterol 150 mg/day; sodium 2,300 mg/day; potassium 4,700 mg/day; calcium 1,250 mg/day; magnesium 500 mg/day; and fiber 30 g/day.
  Other Names: DASH diet
  Arms: Intervention Group
Other: Nutrition education program — The nutrition education program will consist of four lectures intended to improve the overall participants' dietary habits. The lectures will be interactive and will be organized in smaller groups (up to 10 participants) covering the following themes: My Plate dietary guidelines; Principles of a balanced diet; Reading and understanding food nutrition labels; Dietary recommendations for elevated blood pressure, dyslipidemia, and diabetes mellitus.

SUMMARY:
Metabolic syndrome is a term used to describe a complex clinical condition that includes abdominal obesity, increased level of serum triglycerides, elevated blood pressure, decreased level of high-density lipoprotein cholesterol, and high fasting glucose level. Metabolic syndrome represents one of the major risk factors for the development of cardiovascular diseases and type 2 diabetes mellitus. According to the results of numerous previously conducted studies, the prevalence of metabolic syndrome among the individuals with schizophrenia is higher than in the general population.

The reasons for the higher prevalence of metabolic syndrome among the individuals with schizophrenia are not yet fully clarified. Nevertheless, unhealthy dietary habits are considered to be one of the main factors that could have an impact on metabolic syndrome development. According to the results of published studies, individuals with schizophrenia have poorer dietary habits when compared to people without mental disorders.

Although there are numerous previously published studies focused on the impact of nutritional interventions on metabolic syndrome in individuals with schizophrenia, there is still no consensus on what would be the most appropriate nutrition therapy for the treatment of metabolic syndrome in this specific population group. Furthermore, the vast majority of the published studies have been conducted on outpatients, with only a small number of them being carried out on hospitalized individuals with a diagnosis of schizophrenia.

Dietary Approaches to Stop Hypertension (DASH) diet is primarily intended to those individuals with elevated blood pressure, but according to some authors, it could have beneficial effects in the treatment of the metabolic syndrome as well. DASH diet represents a healthy way of eating with a special emphasis on low-fat dairy products, fruits, vegetables and whole grains, together with an overall reduction in sodium intake.

Therefore, the present study aims to determine the impact of dietary habits and nutrition intervention on metabolic syndrome parameters in hospitalized individuals with the diagnosis of schizophrenia.

The investigators hypothesize that the intervention will result in the improvement in metabolic syndrome parameters, the amelioration in dietary habits, and the reduction in body weight.

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis of schizophrenia according to the 10th Revision of the International Classification of Diseases (ICD-10)
* age 18-67
* the diagnosis of metabolic syndrome according to the Joint Interim Statement definition
* taking antipsychotic medication for the last 6 months or more
* a stable phase of schizophrenia
* provided written informed consent (for participants deprived of legal capacity, provided written informed consent of both the participants and their legal guardians)

Exclusion Criteria:

* older than 67
* without the diagnosis of schizophrenia and/or metabolic syndrome
* following one of the specific hospital diets with the restrictions related to the intake of specific food items, groups or nutrients
* taking medications for the reduction of body weight
* significant body weight loss in the past 3 months
* refusing to provide written informed consent
* on personal request
* deterioration in participant's mental state
* the occurrence of a new illness that could unable full participation in the study or could have an interfering effect
* a significant change in pharmacological therapy during the intervention period
* cognitive impairments that unable full participation in the study
* lack of interest or refusal to fully participate in the study
* hospital discharge during the intervention period

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Change in waist circumference | Baseline and after three months
  Waist circumference measuring (in cm) will be performed prior to and immediately after the intervention using a non-strechable measuring tape.
Change in blood pressure | Baseline and after three months
  The assessment of blood pressure (in mmHg) will be performed prior to and immediately after the intervention using an aneroid blood pressure gauge.
Change in high-density lipoprotein cholesterol | Baseline and after three months
  The blood serum concentration of high-density lipoprotein cholesterol (in mmol/L) will be determined prior to and immediately after the intervention. Blood samples will be collected after the overnight fast and the analysis will be performed on the Cobas c 111 analyzer.
Change in serum triglycerides | Baseline and after three months
  The concentration of serum triglycerides (in mmol/L) will be determined prior to and immediately after the intervention. Blood samples will be collected after the overnight fast and the analysis will be performed on the Cobas c 111 analyzer.
Change in fasting blood glucose | Baseline and after three months
  The blood serum concentration of glucose (in mmol/L) will be determined prior to and immediately after the intervention. Blood samples will be collected after the overnight fast and the analysis will be performed on the Cobas c 111 analyzer.

SECONDARY OUTCOMES:
Change in dietary habits | Baseline and after three months
  Dietary habits will be assessed using the nutrition section of Dlugosch & Krieger's General Health Behavior Questionnaire both prior to and immediately after the intervention.
Change in individual food purchase habits | Baseline and after three months
  Individual food purchase diaries, collected at the beginning and at the end of the intervention period, will be used for the evaluation of the changes in individual food purchase habits.
Dietary intake during the intervention | 3 months
  Dietary intake during the intervention will be assessed using three non-consecutive 24-hour dietary recalls (two weekdays and one weekend day).
Change in participants' mental condition | Baseline and after three months
  The global severity of the psychotic illness and severity of specific syndromes within psychotic illness will be evaluated prior to and immediately after the intervention using Signs and Symptoms of Psychotic Illness (SSPI) scale. The scale consists of 20 items (signs and symptoms of psychotic illness). For each item (subscale) a score in the range 0 - 4 is assigned: 0 - no psychopatology; 1 - a deviation questionably pathological; 2 - mild pathological deviation; 3 - pathology of moderate severity; 4 - severe psychopathology. Subscales are summed to determine a global severity of psychotic illness. The highest total score is 80.
Change in body weight | Baseline and after three months
  Body weight (in kg) will be measured prior to and immediately after the intervention using a digital medical scale witl stadiometer.
Change in body mass index | Baseline and after three months
  The measured values of body height and weight will be used for the calculation of body mass index (in kg/m^2).
Change in waist-to-hip ratio | Baseline and after three months
  The waist-to-hip ratio will be calculated from the measured values of waist and hip circumferences: waist circumference (cm) / hip circumference (cm).
Change in body fat percentage | Baseline and after three months
  Determination of body fat percentage will be performed using OMRON BF500 analyzer.
Change in total cholesterol | Baseline and after three months
  The concentration of total cholesterol (in mmol/L) will be determined prior to and immediately after the intervention. Blood samples will be collected after the overnight fast and the analysis will be performed on the Cobas c 111 analyzer.
Change in low-density lipoprotein cholesterol | Baseline and after three months
  The concentration of low-density lipoprotein cholesterol (in mmol/L) will be determined prior to and immediately after the intervention. Blood samples will be collected after the overnight fast and the analysis will be performed on the Cobas c 111 analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Sorić, MSc, Principal Investigator — Psychiatric Hospital Ugljan
Locations (1):
- Psychiatric Hospital Ugljan, Ugljan, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grundy SM, Cleeman JI, Daniels SR, Donato KA, Eckel RH, Franklin BA, Gordon DJ, Krauss RM, Savage PJ, Smith SC Jr, Spertus JA, Costa F; American Heart Association; National Heart, Lung, and Blood Institute. Diagnosis and management of the metabolic syndrome: an American Heart Association/National Heart, Lung, and Blood Institute Scientific Statement. Circulation. 2005 Oct 25;112(17):2735-52. doi: 10.1161/CIRCULATIONAHA.105.169404. Epub 2005 Sep 12. No abstract available. PMID 16157765
- [Background] Xu H, Li X, Adams H, Kubena K, Guo S. Etiology of Metabolic Syndrome and Dietary Intervention. Int J Mol Sci. 2018 Dec 31;20(1):128. doi: 10.3390/ijms20010128. PMID 30602666
- [Background] Vancampfort D, Stubbs B, Mitchell AJ, De Hert M, Wampers M, Ward PB, Rosenbaum S, Correll CU. Risk of metabolic syndrome and its components in people with schizophrenia and related psychotic disorders, bipolar disorder and major depressive disorder: a systematic review and meta-analysis. World Psychiatry. 2015 Oct;14(3):339-47. doi: 10.1002/wps.20252. PMID 26407790
- [Background] Dipasquale S, Pariante CM, Dazzan P, Aguglia E, McGuire P, Mondelli V. The dietary pattern of patients with schizophrenia: a systematic review. J Psychiatr Res. 2013 Feb;47(2):197-207. doi: 10.1016/j.jpsychires.2012.10.005. Epub 2012 Nov 12. PMID 23153955
- [Background] Ratliff JC, Palmese LB, Reutenauer EL, Liskov E, Grilo CM, Tek C. The effect of dietary and physical activity pattern on metabolic profile in individuals with schizophrenia: a cross-sectional study. Compr Psychiatry. 2012 Oct;53(7):1028-33. doi: 10.1016/j.comppsych.2012.02.003. Epub 2012 Mar 16. PMID 22425530
- [Background] Amani R. Is dietary pattern of schizophrenia patients different from healthy subjects? BMC Psychiatry. 2007 May 2;7:15. doi: 10.1186/1471-244X-7-15. PMID 17474979
- [Background] Leao LS, de Moraes MM, de Carvalho GX, Koifman RJ. Nutritional interventions in metabolic syndrome: a systematic review. Arq Bras Cardiol. 2011 Sep;97(3):260-5. doi: 10.1590/s0066-782x2011001200012. English, Portuguese. PMID 22030698
- [Background] Hill AM, Harris Jackson KA, Roussell MA, West SG, Kris-Etherton PM. Type and amount of dietary protein in the treatment of metabolic syndrome: a randomized controlled trial. Am J Clin Nutr. 2015 Oct;102(4):757-70. doi: 10.3945/ajcn.114.104026. Epub 2015 Sep 9. PMID 26354540
- See also: DASH diet description, health benefits and main characteristics — https://www.nhlbi.nih.gov/health-topics/dash-eating-plan